CLINICAL TRIAL: NCT02094300
Title: Zenith® Dissection Endovascular System
Acronym: STABLE I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-622
Record Dates: First submitted 2014-02-21; First posted 2014-03-21 (Estimated); Results first posted 2015-09-14 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-12

CONDITIONS: Aortic Dissection
Keywords: Aorta; Thoracic; Aortic dissection; Rupture; Type B; DeBakey type III; Endovascular
MeSH Terms: conditions — Aortic Dissection; Rupture

ARMS (1):
- Endovascular (Experimental)
  Interventions: Device: Zenith® Dissection Endovascular Graft

INTERVENTIONS:
Device: Zenith® Dissection Endovascular Graft — Instead of making a large incision in the chest, the physician makes a small incision near each hip to insert, and guide the study device(s) into place in the aorta.
  Other Names: Endovascular graft; Stent-graft

SUMMARY:
The Zenith® Dissection Clinical Trial is a clinical trial approved by US FDA to study the safety and effectiveness of the Zenith® Dissection Endovascular System in the treatment of patients with aortic dissection.

ELIGIBILITY:
Inclusion Criteria:

* Branch vessel obstruction/compromise
* Peri-aortic effusion/hematoma
* Resistant hypertension
* Persistent pain/symptoms
* Transaortic growth >5 mm within 3 months
* Transaortic diameter >40 mm.

Exclusion Criteria:

* Age <18 years;
* Other medical condition (e.g., cancer, congestive heart failure) that may cause the patient to be non-compliant with the protocol, confound the results, or is associated with limited life expectancy (i.e., less than 2 years)
* Pregnant, breast-feeding, or planning on becoming pregnant within 24 months;
* Unwilling or unable to comply with the follow-up schedule
* Inability or refusal to give informed consent
* Simultaneously participating in another investigative device or drug study. (The patient must have completed the primary endpoint of any previous study at least 30 days prior to enrollment in this study.)
* Additional medical restrictions as specified in the Clinical Investigation Plan, or
* Additional anatomical restrictions as specified in the Clinical Investigation Plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-12; Primary Completion 2012-02 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Lombardi, MD, Principal Investigator — The Cooper Health System
Locations (5):
- United States (5):
  - University of Florida, Gainesville, Florida
  - Massachusetss General Hospital, Boston, Massachusetts
  - Cooper University Hospital, Camden, New Jersey
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University Hospital, Philadephia, Pennsylvania

REFERENCES:
- [Derived] Lombardi JV, Cambria RP, Nienaber CA, Chiesa R, Mossop P, Haulon S, Zhou Q; STABLE I Investigators. Five-year results from the Study of Thoracic Aortic Type B Dissection Using Endoluminal Repair (STABLE I) study of endovascular treatment of complicated type B aortic dissection using a composite device design. J Vasc Surg. 2019 Oct;70(4):1072-1081.e2. doi: 10.1016/j.jvs.2019.01.089. Epub 2019 May 28. PMID 31147139

RESULTS

PARTICIPANT FLOW:
Groups:
- Zenith® Dissection Endovascular Graft: The Zenith® Dissection Endovascular System is intended for the treatment of patients with aortic dissection of the descending thoracic aorta having anatomy amenable to endovascular repair.
Period: Overall Study
Arm/Group | Zenith® Dissection Endovascular Graft
Started | 26
30 Days | 24
Completed | 6
Not Completed | 20
Not completed — Death | 7
Not completed — Lost to Follow-up | 10
Not completed — Still be eligible for follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Zenith® Dissection Endovascular Graft
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (15)
Gender [Count of Participants; unit: Participants]
  Female | 7
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Major Complications
Description: Major complication is defined as: Retrograde dissection, cardiac events requiring surgical management, prolonged ventilation requiring tracheotomy, renal failure requiring dialysis (where not previously needed), aortic fistula, mesenteric ischemia requiring surgical management, paralysis or paraparesis unresolved after 30 days of therapy, pulmonary embolism, stroke, and multi-system organ failure, unless related to presenting condition.
Time Frame: 30 days
Population: There were 8 patients experienced 30-day major complications.
Measure: Number; unit: participants
Arm/Group | Zenith® Dissection Endovascular Graft
Number analyzed (Participants) | 26
participants
  Paralysis or paraparesis unresolved after 30 days | 2
  Stroke | 4
  Retrograde Type A dissection | 2
  Renal failure requiring dialysis | 3
  Prolonged ventilation requiring tracheotomy | 3

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Zenith® Dissection Endovascular Graft
Serious Adverse Events (participants affected / at risk) | 2/26
Other Adverse Events (participants affected / at risk) | 15/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® Dissection Endovascular Graft (N=26)
Rupture of the aorta at the original entry tear (Vascular disorders) | 1 (1) — Rupture was determined as the cause of death. Site reported that it was related to a pre-existing condition and not the device, clinical events committee (CEC) adjudicated that it was procedure and technique related.
Stroke, midbrain and cerebellar (Nervous system disorders) | 1 (1) — Stroke was determined as the cause of death. clinical events committee (CEC) adjudicated that it was procedure related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® Dissection Endovascular Graft (N=26)
Arrhythmia requiring intervention or new treatment (Cardiac disorders) | 4 (4)
Refractory hypertension (Cardiac disorders) | 3 (3)
Paralytic ileus > 4 days (Gastrointestinal disorders) | 2 (2)
Stroke (Nervous system disorders) | 4 (4)
Pleural effusion requiring treatment (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia requiring antibiotics (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary event requiring tracheostomy or chest tube (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Ventilation > 24 hours (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Renal failure requiring dialysis (Renal and urinary disorders) | 3 (3)
Serum creatinine rise > 30% above baseline resulting in a persistent value > 2.0 mg/dl (Renal and urinary disorders) | 3 (3)
Post-procedure transfusion (Vascular disorders) | 7 (9)
Vascular injury (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days